CLINICAL TRIAL: NCT02966158
Title: A Randomized Controlled Trial in Women With Coronary Artery Disease Investigating the Effects of Aerobic Interval Training Versus Moderate Intensity Continuous Exercise in the Standard Cardiac Rehabilitation Setting: Aerobic Exercise Capacity and Cognitive Function
Brief Title: A Randomized Controlled Trial in Women With Coronary Artery Disease Investigating the Effects of Aerobic Interval Training Versus Moderate Intensity Continuous Exercise
Acronym: CAT vs MICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Paul Oh, Medical Director, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-5900
Record Dates: First submitted 2016-10-13; First posted 2016-11-17 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Coronary Artery Disease
Keywords: Aerobic Interval Training; Fitness; Endothelial Function; Cognition
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIT Group (Experimental): The AIT Group will perform usual care CR exercise for the 1st month of the program. This includes performing aerobic exercise 5 times/week and resistance training twice/week (offered 2 weeks after program start). In month two, this group will begin to perform AIT three days/week, along with two MICE and two RT sessions.
  The AIT exercise protocol includes the following components:
  1. Warm Up Period: 5-10 minutes of walking performed at an intensity that will feel fairly light. Heart rate monitors and watches will be used to gauge their effort.
  2. Intervals: Between two to four 4-minute intervals of walking/jogging performed at an intensity that is close to participants' maximal effort, based on the exercise tests that were performed at the beginning of the program. These "hard intervals" will be separated by 3-minutes of active recovery performed at a very light intensity.
  3. Cool Down Period: 5 minutes of walking performed at a fairly light intensity.
  Interventions: Other: AIT Group
- MICE Group (No Intervention): This group will perform usual care CR for 6 months, which includes both resistance and aerobic exercise (MICE) training. Aerobic exercise is prescribed in the first exercise class and performed 5 times/week, the resistance training program is offered after 2 weeks in the program and performed 2 times/week. Participants will be asked to keep a record of the exercise that they do.
  Resistance/Strength Training: Patients will be performing 1-2 sets of 5 to 10 resistance training exercises using a combination of hand-held dumbbells, elastic bands of varying thicknesses, as well as their own body weight for resistance.
  Aerobic Training: Patients will have their aerobic exercise prescription set at an intensity and duration that will be comfortable for them, based on the tests conducted at the beginning of the program to ensure their safety.

INTERVENTIONS:
Other: AIT Group — The AIT Group will begin with a one-month, "run-in" period where patients will perform current standard of care CR programming, which will involve traditional MICE. MICE at the Cardiac Rumsey Centre will consist of either track walking/jogging or treadmill walking/jogging for approximately 30-40 minutes, performed at an intensity of 60-80% of VO2peak, in addition to a warm-up and cool down period. In the second month of the study intervention, patients will begin to perform AIT three days per week, which involves performing 4-minute intervals at greater than 90% of peak heart rate, separated by 3-minutes of active recovery, with one of those AIT exercise sessions occurring at the Rumsey Centre under supervision, and 2 sessions per week of MICE, which will again consist of the 30-40 minutes of walking/jogging at an intensity of 60-80% of VO2peak, with an allotted warm up and cool down period.
  Other Names: Aerobic Interval Training Intervention Group
  Arms: AIT Group

SUMMARY:
Heart disease is the number one killer amongst chronic diseases around the world, and it is responsible for taking the lives of an estimated 17.5 million people each year. Exercise-based cardiac rehabilitation (CR) programs, which help heart patients improve their current health, prevent future heart problems, and improve their quality of life, are an effective strategy for lowering the risk of heart-related deaths in heart patients. CR programs currently have their patients perform moderate intensity, continuous exercise (MICE), which traditionally takes the form of walking, jogging, or cycling at a comfortable pace for 30-60 minutes. Recently, aerobic interval training (AIT), which involves performing short bouts of exercise, typically ranging from 15 seconds to four minutes at near maximal effort, followed by periods of recovery or rest, has emerged as a more effective strategy than MICE for lowering the risk of heart-related deaths in heart patients. Although these initial findings appear to hold much promise for improving CR programs in the future, it is important to recognize that women have been underrepresented or not included in these studies to date. Therefore, the goal of this study is to determine the effects of AIT versus MICE on the risk of heart-related death, blood vessel health, and brain health in women who have heart disease, and who have been referred to a six-month, outpatient CR program.

DETAILED DESCRIPTION:
This will be the first randomized controlled trial (RCT) investigating the effects of AIT versus MICE on aerobic exercise capacity, endothelial function, and cognition, in women only, who have CAD and have been referred to the six-month, outpatient CR program at the Toronto Rehabilitation Institute (TRI)-Cardiac Rumsey Centre. Study participants will be reporting to the Rumsey Centre one day per week for a combination of supervised exercise sessions and educational seminars or workshops, and they will be performing four additional unsupervised, home-exercise sessions per week for a target total of five exercise sessions per week.

Recruitment and Sampling

Immediately after completion of a symptom-limited intake CPA, a previously identified eligible patient who would have been screened for eligibility upon her referral to the six-month, outpatient CR program at the TRI-Cardiac Rumsey Centre will be asked by either the Cardiopulmonary Exercise Technicians, or Lab Coordinator performing the initial CPA, if she would be interested in speaking to a researcher and learning more about potential participation in this research study. If the patient agrees to speak to the researcher, the researcher will meet the patient in person immediately following the CPA to explain the study and to obtain voluntary, written and informed consent if applicable. Patients will be provided with the opportunity to take the consent forms home, and to discuss participation in the study with their spouses or other family members, etc., and to take as much time is required to decide whether participation in the study is a desirable option for them.

If, and when a patient provides written and informed consent to participate in the study, she will be randomized by a computerized random number generator (operated by a blinded third party researcher) to either the six-month standard of care CR program offered at the TRI-Rumsey Centre involving MICE, or to the 6-month AIT intervention. Both the MICE and AIT arms of the study will consist of patients attending one, supervised exercise session per week at the TRI-Rumsey Centre, and they will perform four additional unsupervised home-exercise sessions per week for a total of five exercise sessions per week as the goal.

The AIT Intervention

The AIT Group will begin with a one-month, "run-in" period where patients will perform current standard of care CR programming, which will involve traditional MICE. MICE at the Cardiac Rumsey Centre will consist of either track walking/jogging or treadmill walking/jogging for approximately 30-40 minutes, performed at an intensity of 60-80% of VO2peak, in addition to a warm-up and cool down period. In the second month of the study intervention, patients will begin to perform AIT three days per week, with one of those AIT exercise sessions occurring at the Rumsey Centre under supervision, and 2 sessions per week of MICE, which will again consist of the 30-40 minutes of walking/jogging at an intensity of 60-80% of VO2peak, with an allotted warm up and cool down period.

The AIT Exercise Protocol

Upon examination of the most recent RCTs investigating AIT versus MICE between 2004 and 2016, specifically in the CAD population, the AIT intervention group experienced greater improvements in VO2peak, which translated to ~1.5-2 mL kg-1 min-1 improvements compared to the MICE (control) group. These results are compelling, particularly in the context of a potential 10-25% reduction in cardiovascular mortality risk above and beyond what would have been conferred by standard of care MICE prescription. In almost 90% of these most recent RCTs comparing the effects of AIT versus MICE on aerobic exercise capacity in CAD patients, the AIT exercise protocol consisted of 4x4 minute intervals of treadmill walking at either 80-90% of VO2peak, or 85-95% of HRpeak, or 80-90% of Heart Rate Reserve (HRR=HRpeak-resting HR), with 3 minutes of active recovery between the 4-minute intervals, performed at an intensity of ~50-70% of VO2peak, HRpeak, or HRR.

Therefore, in remaining consistent with the previous literature supporting AIT in CAD patients, the AIT exercise protocol that the participants will be executing in this study consists of the following components:

1. Warm Up Period: 5-10 minutes of walking performed at 50%-60% of VO2peak and/or the corresponding HR (~60%-70% HRpk) and/or RPE of ~10-12 on the Borg Scale
2. Intervals: Four 4-minute intervals of walking/jogging performed at an intensity of 85-95% of VO2peak, or >90% of HRpk, and/or RPE >17 on the Borg Scale, interspersed with 3-minutes of active recovery performed at an intensity of ~50%-70% HRpk
3. Cool Down Period: 5 minutes of walking performed at an intensity of 50-70% HRpk, and/or RPE ~10-12 on the Borg Scale Understanding that we must be cognizant of the fact that each study participant may respond and progress to this AIT intervention at different rates, it is our intention to begin with two 4-minute intervals in the first week of the AIT intervention, and then to progress participants to performing three, and then eventually four 4-minute intervals by the fourth week of the intervention, i.e. the end of Month 2 in the study/CR program timeline. The decision to progress patients accordingly will be made judiciously upon deliberation of both researcher and cardiac rehabilitation supervisor/case manager for each study participant.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with CAD
* In sinus rhythm
* Left Ventricular Ejection fraction>35%
* >3 weeks post myocardial infarction (MI) or percutaneous intervention (PCI)
* >4 weeks post coronary artery bypass graft (CABG)
* Ability to provide written and informed consent

Exclusion Criteria:

* Any major musculoskeletal, pulmonary, or psychiatric comorbidity that precludes participation in aerobic and resistance training exercise
* Canadian Cardiovascular Society (CCS) contraindications that present upon initial intake Cardiopulmonary Exercise Assessment (CPA), which include Class II-IV angina, significant arrhythmia, or >1mm horizontal/downsloping ST-segment depression.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Aerobic Exercise Capacity | Change from baseline aerobic exercise capacity at 6 months
  Aerobic exercise capacity, as measured directly by VO2peak, will be measured via breath-by-breath gas exchange analysis captured by a metabolic cart (Vmax Encore, SensorMedics, Yorba Linda, CA), while a patient is performing a symptom-limited CPA using a cycle ergometer (Ergoselect 200P, Ergoline, Bitz, Germany).
Cognitive Function | Change from baseline cognitive function at 6 months
  A battery of neuropsychological tests were chosen to assess cognitive function based on harmonized standards in accordance with the National Institute of Neurological Disorders and Stroke and Canadian Stroke Network [32].

SECONDARY OUTCOMES:
Endothelial Function | Baseline, 3 months, and 6 months
  Blood vessel health is assessed by the change in flow-mediated dilation of the brachial artery.
Quality of Life | Baseline and 6 months
  Standard cardiac rehab medical health questionnaire will be used to capture quality of life.
Cardiovascular Risk Profile | Baseline and 6 months
  This will be assessed by standard blood requisition blood draw capturing lipid, cholesterol, and triglyceride levels, in addition to the measurement of anthropometrics, such as height, body mass, waist circumference, and systolic and diastolic blood pressure values.
Adherence to Exercise | Throughout 6 month exercise program
  Adherence to the exercise interventions will be captured by HR and speed data uploaded and analyzed using the Garmin Forerunner 620 GPS watch (Garmin, Olathe, KS, USA) and accompanying heart rate monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Paul I Oh, MD, MSc, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network Cardiac Rumsey Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data IPD will be shared with other researchers upon request (i.e. contacting researchers via email, phone, etc,.) once the study is complete and the data is shared and presented through publication. IPD may be used for secondary purposes, such as in meta-analyses, or in re-analyses including different comparator groups, and for the replication of results.

REFERENCES:
- [Derived] Lee LS, Tsai MC, Brooks D, Oh PI. Randomised controlled trial in women with coronary artery disease investigating the effects of aerobic interval training versus moderate intensity continuous exercise in cardiac rehabilitation: CAT versus MICE study. BMJ Open Sport Exerc Med. 2019 Oct 22;5(1):e000589. doi: 10.1136/bmjsem-2019-000589. eCollection 2019. PMID 31749981